CLINICAL TRIAL: NCT01054027
Title: A Randomized Controlled Trial to Determine the Lowest Effective Dose for Adequate Mydriasis in Premature Infants
Brief Title: Study on Effective Mydriasis in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Monisha Bahri, Georgetown University Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: 2007-109
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Retinopathy of Prematurity (ROP)
Keywords: Retinopathy of Prematurity (ROP); Eye exams; Premature infants; cyclomydril
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth | interventions — Phenylephrine; Cyclopentolate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0 Drop (Experimental): Left eye dose
  Interventions: Drug: 1% phenylephrine and 0.2% cyclopentolate
- 1 Drop (Experimental): Left eye dose
  Interventions: Drug: 1% phenylephrine and 0.2% cyclopentolate
- 2 drop (Experimental): Left eye dose
  Interventions: Drug: 1% phenylephrine and 0.2% cyclopentolate
- 3 drops (Active Comparator): Right eye dose for all groups
  Interventions: Drug: 1% phenylephrine and 0.2% cyclopentolate

INTERVENTIONS:
Drug: 1% phenylephrine and 0.2% cyclopentolate — given as drops, prior to eye exam
  Other Names: Cyclomydril

SUMMARY:
The purpose of this study is to compare the dilating effect of 0, 1, 2 or 3 drops of mydriatic (pupil dilating) in premature infants undergoing routine retinal (eye) screening exams for Retinopathy of Prematurity (ROP).

DETAILED DESCRIPTION:
Premature infants need to have eye exams starting at about 4 weeks of age and continuing until their retinas (membrane at the back of the eye which collects and transfers light) is fully grown. These exams are done to see if they have developed ROP, a disease which can lead to blindness if not treated.

The ophthalmologist (eye doctor) looks through the enlarged pupil (opening at the front of the eye) to see the retina. The drug that is used to dilate the pupil, Cyclomydril, has been shown to have side effects in premature infants. No literature has shown what the optimal dose is for premature babies. Nursery policy is to give 3 drops of Cyclomydril in each eye, at 5 minute intervals, 45-60 minutes before a scheduled eye exam. We sought to reduce the dose without delaying the exam for an under-sized pupil.

In the study, each infant is randomized at the time of the exam to receive either 0, 1 or 2 drops of Cyclomydril in the left eye and 3 drops in the right eye to serve as their own control. The zero-drop group was created to test the contralateral (opposite eye) effect of 3 drops in the right eye. Pupil dilation size is measured using the Colvard pupillometer by a Pediatric Ophthalmologist examiner (G.V.V.) who was not masked to study group assignment.

Measures of pupil size are done at baseline (before any drops given), 45, 90 and 120 minutes after the first drop was given. ROP screening exam is done at the first opportunity to visualize the posterior and peripheral retina.

Additional drops are given at 120 minutes if the observer is unable to complete the exam prior to that point.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants undergoing clinically indicated retinal exams

Exclusion Criteria:

* Ocular congenital anomalies
* Pre-threshold ROP

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-03; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
dilation of the pupil in millimeters | at baseline (no drops yet instilled), 45, 90 and 120 minutes after drops instilled

CONTACTS AND LOCATIONS:
Overall Officials: Monisha Bahri, MD, Principal Investigator — Georgetown University Hospital
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States